CLINICAL TRIAL: NCT04222387
Title: Investigation of Potential Retinal Toxicity Associated With Hair Dye Products Containing pPD (Para-phenylenediamine) Type Aromatic Amines
Brief Title: Investigation of Potential Retinal Toxicity Associated With Hair Dye Products Containing pPD Type Aromatic Amines
Acronym: CAPITOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CSA_2019_13
Record Dates: First submitted 2019-12-11; First posted 2020-01-10 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: MEK Inhibitor-Associated Serous Retinopathy
Keywords: MEK Inhibitor-Associated Serous Retinopathy; Hair dye; Aromatic amines

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with hair dye (Experimental): Hair dye product with pPD Type Aromatic Amines used up to 1 month before
  Interventions: Device: OCT-B scan

INTERVENTIONS:
Device: OCT-B scan — OCT-B scan (Optical coherence tomography)

SUMMARY:
Hair dye products could induce minimal forms of MEKAR retinopathies (Mitogen-activated Extracellular signal-regulated Kinase - inhibitors associated retinopathies). These minimal forms of MEKAR are likely to be underdiagnosed, since the associated visual loss is usually mild and so this condition should be considered when patients report blurred vision. The aim of the study is to analyze whether in the current population that dyes the hair, minimal forms that go unnoticed by MEKAR retinopathies can be induced.

ELIGIBILITY:
Inclusion Criteria:

* Hair dye up to one month before the inclusion
* Hair dye product containing aromatic amines

Exclusion Criteria:

* Pregnant or lactating woman
* Retinal pathology already known, or central serous choroiditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
% of patients with MEKAR retinopathy detected on OCT-B scan | Day of inclusion, up to one month month after the last hair dye
  Physiological parameter : Serous retinal detachment at the posterior pole, detected on OCT-B scan

CONTACTS AND LOCATIONS:
Overall Officials: Claire SCEMAMA, MD, Principal Investigator — cstimsit@for.paris
Locations (1):
- Fondation A de Rothschild, Paris, France